CLINICAL TRIAL: NCT00001337
Title: Dose-Adjusted EPOCH Chemotherapy and Rituximab (CD20+) in Adults and Children With Previously Untreated Patients With Aggressive Non-Hodgkin's Lymphoma
Brief Title: Dose-Adjusted EPOCH Chemotherapy and Rituximab (CD20+) in Previously Untreated Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Roschewski, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 930133; 93-C-0133; NCT00018980 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL); Primary Mediastinal Large B-cell Lymphoma; Burkitt Lymphoma; Anaplastic Large-Cell Lymphoma; Gray Zone Lymphoma
Keywords: Primary Mediastinal B-Cell Lymphoma; CD20 +; Diffuse Large B-Cell Lymphoma; Anaplastic Large Cell Lymphoma; De Novo
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Etoposide; Rituximab; Prednisone; Cyclophosphamide; Vincristine; Doxorubicin; liposomal doxorubicin; Magnetic Resonance Imaging; Tomography, X-Ray Computed; Biopsy; Positron-Emission Tomography; Laparotomy; Ondansetron; Prochlorperazine; Omeprazole; omeprazole, sodium bicarbonate drug combination; Dioctyl Sulfosuccinic Acid; Sennosides; doxidan; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) (Experimental): Subgroup 1 (SG1) - All participants who received combination Rituximab (EPOCH-R). Rituximab 375 mg/m^2 intravenous (IV) on day 1, every 21 days, prednisone 100mg by mouth (PO) twice a day (bid) on days 1 through 5 every 21 days, and cyclophosphamide 750mg/m^2 on day 5 every 21 days. Doxorubicin 10mg/m^2/day, vincristine 0.4mg/m^2/day, and etoposide 50mg/m^2/day were delivered as continuous intravenous (CIV) infusions over 96 hours starting on day 1 every 21 days. Dose levels were adjusted on doxorubicin, etoposide, and cyclophosphamide each cycle based on neutrophil nadir.
  Interventions: Drug: Etoposide; Biological: Rituximab; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Diagnostic Test: MRI; Diagnostic Test: CT; Procedure: Biopsy; Diagnostic Test: PET scan; Procedure: Laparotomy; Other: Ondansetron; Other: Prochlorperazine; Other: Omeprazole; Other: Docusate Sodium + Sennosides; Other: Lactulose
- EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide) (Experimental): Subgroup 2 (SG2) - EPOCH alone: All participants who received Prednisone 100mg by mouth (PO) twice a day (bid) on days 1 through 5 every 21 days, and cyclophosphamide 750mg/m^2 on day 5 every 21 days. Doxorubicin 10mg/m^2/day, vincristine 0.4mg/m^2/day, and etoposide 50mg/m^2/day were delivered as continuous intravenous (CIV) infusions over 96 hours starting on day 1 every 21 days. Dose levels were adjusted on doxorubicin, etoposide, and cyclophosphamide each cycle based on neutrophil nadir.
  Interventions: Drug: Etoposide; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Diagnostic Test: MRI; Diagnostic Test: CT; Procedure: Biopsy; Diagnostic Test: PET scan; Procedure: Laparotomy; Other: Ondansetron; Other: Prochlorperazine; Other: Omeprazole; Other: Docusate Sodium + Sennosides; Other: Lactulose

INTERVENTIONS:
Drug: Etoposide — Etoposide 50mg/m^2/day were delivered as continuous intravenous (CIV) infusions over 96 hours starting on day 1 every 21 days.
  Combination chemotherapy given with Rituximab, Etoposide, VP-16; Prednisone, Cyclophosphamide, Vincristine, and Doxorubicin (EPOCH-R) intravenous (IV) every 3 weeks for 6 cycles.
  Other Names: VP-16
Biological: Rituximab — Rituximab given on Day 1 of combination chemotherapy (EPOCH-R) every 3 weeks for 6 cycles.
  Combination chemotherapy given with Rituximab, Etoposide, VP-16; Prednisone, Cyclophosphamide, Vincristine, and Doxorubicin (EPOCH-R) intravenous (IV) every 3 weeks for 6 cycles.
  Other Names: Rituxan
  Arms: With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab)
Drug: Prednisone — Prednisone 100mg by mouth (PO) twice a day (bid) on days 1 through 5 every 21 days.
  Combination chemotherapy given with Rituximab, Etoposide, VP-16; Prednisone, Cyclophosphamide, Vincristine, and Doxorubicin (EPOCH-R) intravenous (IV) every 3 weeks for 6 cycles.
  Other Names: Rayos; Deltasone; Prednisone Intensol
Drug: Cyclophosphamide — Cyclophosphamide 750mg/m^2 on day 5 every 21 days.
  Combination chemotherapy given with Rituximab, Etoposide, VP-16; Prednisone, Cyclophosphamide, Vincristine, and Doxorubicin (EPOCH-R) intravenous (IV) every 3 weeks for 6 cycles.
  Other Names: Cytoxan
Drug: Vincristine — Vincristine 0.4mg/m^2/day.
  Combination chemotherapy given with Rituximab, Etoposide, VP-16; Prednisone, Cyclophosphamide, Vincristine, and Doxorubicin (EPOCH-R) intravenous (IV) every 3 weeks for 6 cycles.
  Other Names: Marqibo; Vincasar PFS
Drug: Doxorubicin — Doxorubicin 10mg/m^2/day.
  Combination chemotherapy given with Rituximab, Etoposide, VP-16; Prednisone, Cyclophosphamide, Vincristine, and Doxorubicin (EPOCH-R) intravenous (IV) every 3 weeks for 6 cycles.
  Other Names: Lipodox; Lipodox 50; Doxil
Diagnostic Test: MRI — Baseline and/or on completion of therapy.
  Other Names: Magnetic resonance imaging
Diagnostic Test: CT — Baseline and/or on completion of therapy.
  Other Names: Computed tomography
Procedure: Biopsy — Baseline and/or on completion of therapy.
Diagnostic Test: PET scan — As clinically indicated.
  Other Names: positron emission tomography scan
Procedure: Laparotomy — As clinically indicated.
Other: Ondansetron — Nausea and/or vomiting.
  Other Names: Zofran ODT; Zuplenz; Zofran
Other: Prochlorperazine — Nausea and/or vomiting.
  Other Names: Compro
Other: Omeprazole — Gastroesophageal reflux disease (GERD).
  Other Names: Prilosec OTC; Zegerid; OmePPi
Other: Docusate Sodium + Sennosides — Constipation.
  Other Names: Senna-Plus; Colace 2-in-1; Dok Plus
Other: Lactulose — Constipation
  Other Names: Kristalose; Enulose; Generlac

SUMMARY:
5-Drug Combination Chemotherapy with Hematologic Toxicity Attenuation. Etoposide phosphate, prednisone, vincristine sulfate (Oncovin), cyclophosphamide, and doxorubicin hydrochloride (hydroxydaunorubicin)(EPOCH): Etoposide, VP-16, NSC-141540; Prednisone, PRED, NSC-10023; Vincristine, VCR, NSC-67574; Cyclophosphamide, CTX, NSC-26271; Doxorubicin, DOX, NSC-123127; with Granulocyte Colony-Stimulating Factor (Amgen), Granulocyte colony-stimulating factor (G-CSF), NSC-614629.

DETAILED DESCRIPTION:
Background:

The treatment of the intermediate and aggressive non-Hodgkin's lymphomas in adults and children commonly induces complete responses in a sizable fraction of the treated population, and about 2/3 of the complete responders appear to have prolonged disease-free survival.

The present study assesses the activity and tolerability in previously untreated patients of a regimen of etoposide phosphate, prednisone, vincristine sulfate (Oncovin), cyclophosphamide, and doxorubicin hydrochloride (hydroxydaunorubicin)(EPOCH) infusional chemotherapy given intensively with granulocyte colony-stimulating factor (G-CSF) support.

Objectives:

Primary:

Assess complete response (CR) and progression-free survival (PFS) of dose-adjusted EPOCH-Rituximab (DA-EPOCH-R) with G-CSF in aggressive B-cell lymphomas.

Eligibility:

Non-Hodgkin's lymphomas in the following categories: mediastinal gray zone lymphoma (MGZL) and primary mediastinal B cell lymphoma (PMBL).

Patients greater than or equal to 12 years old.

Any Stage for PMBL and MGZL.

No prior systemic chemotherapy.

Human immunodeficiency virus (HIV) negative.

Design:

This study will estimate the complete response rate of a group of previously untreated patients and the extent to which EPOCH infusional drug delivery accompanied by a hematopoietic growth factor can increase the dose intensity of treatment.

Patients receive prednisone orally for 5 days, a 96-hour infusion of vincristine, doxorubicin, and etoposide, and a bolus of cyclophosphamide on day 5.

Cycles are repeated every 21 days for a total of 6-8 cycles.

Patients with cluster of differentiation 20 (CD20) expressing tumors (i.e., mature B-cell lymphomas) will also receive rituximab, the humanized monoclonal antibody against the CD20 receptor on day 1 of each cycle.

A total of 348 patients will be enrolled on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Non-Hodgkin's lymphomas in the following categories: mediastinal gray zone lymphoma and primary mediastinal B cell lymphoma.

Diagnosis confirmed by staff of the Hematopathology Section, Laboratory of Pathology, National Cancer Institute (NCI). Tissue blocks from patients treated in extramural sites must be forwarded to the NCI for analysis of B-cell leukemia/lymphoma 2 (bcl-2) by immunohistochemistry (IHC) and other markers within 1 month of study entry.

Patients greater than or equal to 12 years old.

Stage and Prognosis of Patients: Any stage for mediastinal gray zone lymphoma (MGZL) and primary mediastinal B-cell lymphoma (PMBL).

No prior systemic chemotherapy. Patients may be entered if they have had prior limited-field radiotherapy, a short course of glucocorticoids and/or cyclophosphamide for an urgent problem at diagnosis (e.g. epidural cord compression, superior vena cava syndrome).

Human immunodeficiency virus (HIV) negative.

Not pregnant or nursing.

Adequate major organ function [in adults: serum creatinine less than or equal to 1.5 mg/dl or creatinine clearance greater than 60 ml/min; and in children serum creatinine (CR) less than or equal to age-adjusted normal (age 12 to 15 maximum serum creatinine 1.2 mg/dl and age greater than 15 maximum serum creatinine 1.5 mg/dl); bilirubin less than 1.5 mg/dl; absolute neutrophil count (ANC) greater than 1,000 and platelets greater than 100,000) unless impairment is due to organ involvement by lymphoma or immune-mediated mechanism caused by lymphoma.

No active symptomatic ischemic heart disease, myocardial infarction or congestive heart failure within the past year. If multi-gated acquisition (MUGA) is obtained, the left ventricular ejection fraction (LVEF) should exceed 40%.

No other serious concomitant medical illnesses or uncontrolled active infection that would jeopardize the patient's ability to receive the regimen with reasonable safety.

No history of unrelated (non-lymphomatous) neoplasms within past 5 years other than non-melanoma skin cancer or in-situ cancer.

Ability to give informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 1993-05-08 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Holy Cross Hospital, Fort Lauderdale, Fort Lauderdale, Florida
  - University of Maryland, Baltimore, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Luke's Roosevelt Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Klimo P, Connors JM. MACOP-B chemotherapy for the treatment of diffuse large-cell lymphoma. Ann Intern Med. 1985 May;102(5):596-602. doi: 10.7326/0003-4819-102-5-596. PMID 2580468
- [Background] Lai GM, Chen YN, Mickley LA, Fojo AT, Bates SE. P-glycoprotein expression and schedule dependence of adriamycin cytotoxicity in human colon carcinoma cell lines. Int J Cancer. 1991 Nov 11;49(5):696-703. doi: 10.1002/ijc.2910490512. PMID 1682280
- [Background] DeVita VT Jr, Canellos GP, Chabner B, Schein P, Hubbard SP, Young RC. Advanced diffuse histiocytic lymphoma, a potentially curable disease. Lancet. 1975 Feb 1;1(7901):248-50. doi: 10.1016/s0140-6736(75)91142-3. PMID 46388
- [Derived] Lai C, Cole DE, Steinberg SM, Lucas N, Dombi E, Melani C, Roschewski M, Balis F, Widemann BC, Wilson WH. Doxorubicin pharmacokinetics and toxicity in patients with aggressive lymphoma and hepatic impairment. Blood Adv. 2023 Feb 28;7(4):529-532. doi: 10.1182/bloodadvances.2022007431. PMID 35882475
- [Derived] Miljkovic MD, Melani C, Pittaluga S, Lakhotia R, Lucas N, Jacob A, Yusko E, Jaffe ES, Wilson WH, Roschewski M. Next-generation sequencing-based monitoring of circulating tumor DNA reveals clonotypic heterogeneity in untreated PTCL. Blood Adv. 2021 Oct 26;5(20):4198-4210. doi: 10.1182/bloodadvances.2020003679. PMID 34432874
- [Derived] Kurtz DM, Scherer F, Jin MC, Soo J, Craig AFM, Esfahani MS, Chabon JJ, Stehr H, Liu CL, Tibshirani R, Maeda LS, Gupta NK, Khodadoust MS, Advani RH, Levy R, Newman AM, Duhrsen U, Huttmann A, Meignan M, Casasnovas RO, Westin JR, Roschewski M, Wilson WH, Gaidano G, Rossi D, Diehn M, Alizadeh AA. Circulating Tumor DNA Measurements As Early Outcome Predictors in Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2018 Oct 1;36(28):2845-2853. doi: 10.1200/JCO.2018.78.5246. Epub 2018 Aug 20. PMID 30125215
- [Derived] Melani C, Advani R, Roschewski M, Walters KM, Chen CC, Baratto L, Ahlman MA, Miljkovic MD, Steinberg SM, Lam J, Shovlin M, Dunleavy K, Pittaluga S, Jaffe ES, Wilson WH. End-of-treatment and serial PET imaging in primary mediastinal B-cell lymphoma following dose-adjusted EPOCH-R: a paradigm shift in clinical decision making. Haematologica. 2018 Aug;103(8):1337-1344. doi: 10.3324/haematol.2018.192492. Epub 2018 May 10. PMID 29748435
- [Derived] Wilson WH, Pittaluga S, Nicolae A, Camphausen K, Shovlin M, Steinberg SM, Roschewski M, Staudt LM, Jaffe ES, Dunleavy K. A prospective study of mediastinal gray-zone lymphoma. Blood. 2014 Sep 4;124(10):1563-9. doi: 10.1182/blood-2014-03-564906. Epub 2014 Jul 14. PMID 25024303
- [Derived] Dunleavy K, Pittaluga S, Shovlin M, Steinberg SM, Cole D, Grant C, Widemann B, Staudt LM, Jaffe ES, Little RF, Wilson WH. Low-intensity therapy in adults with Burkitt's lymphoma. N Engl J Med. 2013 Nov 14;369(20):1915-25. doi: 10.1056/NEJMoa1308392. PMID 24224624
- [Derived] Dunleavy K, Pittaluga S, Maeda LS, Advani R, Chen CC, Hessler J, Steinberg SM, Grant C, Wright G, Varma G, Staudt LM, Jaffe ES, Wilson WH. Dose-adjusted EPOCH-rituximab therapy in primary mediastinal B-cell lymphoma. N Engl J Med. 2013 Apr 11;368(15):1408-16. doi: 10.1056/NEJMoa1214561. PMID 23574119
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1993-C-0133.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled But Not Treated: One participant was enrolled and not treated.
Period: Overall Study
Arm/Group | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide) | Enrolled But Not Treated
Started | 235 | 112 | 1
Follow-up Period Completed | 148 | 43 | 0
Completed | 148 | 43 | 0
Not Completed | 87 | 69 | 1
Not completed — Switched to alternate treatment | 2 | 2 | 0
Not completed — Refused further treatment | 2 | 1 | 0
Not completed — Began other Tx | 1 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0
Not completed — Doesn't have NHL | 0 | 1 | 0
Not completed — Non protocol tx needed | 3 | 1 | 0
Not completed — Protocol change | 1 | 0 | 0
Not completed — 2nd primary disease | 0 | 0 | 1
Not completed — Death during follow up period | 9 | 4 | 0
Not completed — Death on study | 19 | 9 | 0
Not completed — Disease progression during follow-up period | 3 | 1 | 0
Not completed — Disease progression on study | 33 | 41 | 0
Not completed — Lost to further follow-up | 10 | 6 | 0
Not completed — 2nd malignancy | 1 | 0 | 0
Not completed — Treatment for second lymphoma | 0 | 1 | 0
Not completed — Transfer to transplant | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Collected baseline data is reported for 1 participant enrolled but not treated.
Groups:
- Enrolled But Not Treated: Participant was enrolled but not treated.
- Total: Total of all reporting groups
Arm/Group | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide) | Enrolled But Not Treated | Total
Number analyzed (Participants) | 235 | 112 | 1 | 348
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 0 | 0 | 5
  Between 18 and 65 years | 200 | 102 | 1 | 303
  >=65 years | 30 | 10 | 0 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.97 (17.7) | 47.2 (15.29) | 62.6 (0) | 45.06 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 50 | 0 | 153
  Male | 132 | 62 | 1 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 1 | 0 | 18
  Not Hispanic or Latino | 211 | 108 | 1 | 320
  Unknown or Not Reported | 7 | 3 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 6 | 0 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 37 | 13 | 1 | 51
  White | 169 | 91 | 0 | 260
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 17 | 2 | 0 | 19
Region of Enrollment [Number; unit: participants]
  United States | 235 | 112 | 1 | 348

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (Complete Response + Partial Response)
Description: Overall response defined as a Complete Response + Partial Response was measured by the Response Criteria. Complete Response is disappearance of all signs and symptoms of lymphoma for a period of at least one month. Partial Response is 50% or greater decrease in the sum of the products of the longest perpendicular diameters of all measured lesions lasting for a period of at least one month.
Time Frame: Time frame was from beginning of therapy until the end of therapy, an average of 6 months
Population: 347/348 participants were analyzed because 1 was inevaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide)
Number analyzed (Participants) | 235 | 112
Participants | 216 | 94

2. Primary Outcome: Progression Free Survival (PFS)
Description: The Dixon-Simon method will be used to determine whether large B-cell lymphomas expressing BCL-2 (+) participants may experience an improved progression free survival with Etoposide, VP-16, and Doxorubicin with Prednisone, Cyclophosphamide, and Rituximab (EPOCH-R) compared to EPOCH alone, and to obtain a concurrent, precisely determined measure of progression free survival. PFS is the time from start of treatment to documented evidence of disease progression. Progression is an increase of 25% or more in the sum of the products of the longest perpendicular diameters of all measured lesions, or the appearance of any new lesions measured by the Response Criteria.
Time Frame: Progression free survival was calculated from study entry until progression or death from any cause. Median follow up of evaluable participants was 5 years (range 2-7 years)
Population: 347/348 participants were analyzed because 1 was inevaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide)
Number analyzed (Participants) | 235 | 112
Participants | 73 | 41

3. Secondary Outcome: Proportion of Participants With Serious and/or Non-serious Adverse Events Leading to Discontinuation of Therapy
Description: Here is the proportion of participants with adverse events leading to discontinuation of therapy. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the participant and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Initiation of study drug until 30 days after treatment, an average of 6 months
Population: 347/348 participants were analyzed because one participant was enrolled and not treated.
Measure: Number; unit: proportion of participants
Arm/Group | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide)
Number analyzed (Participants) | 235 | 112
proportion of participants | 0.03 | 0.04

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Time frame is from study entry until 30 days after completing study therapy, approximately 5 years.
Population: 347/348 participants were analyzed because one participant was enrolled and not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide)
Number analyzed (Participants) | 235 | 112
Participants | 235 | 112

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were monitored/assessed from the first study intervention, Study Day 1, through 30 days after the last study intervention was administered, approximately 5 years.
Description: 347/348 participants were analyzed because one participant was enrolled and not treated.
Arm/Group | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide)
All-Cause Mortality (participants affected / at risk) | 28/235 | 13/112
Serious Adverse Events (participants affected / at risk) | 146/235 | 44/112
Other Adverse Events (participants affected / at risk) | 235/235 | 112/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) (N=235) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide) (N=112)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (3) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (7) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cytokine release syndrome/acute infusion reaction (General disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Infections and infestations) | 104 (170) | 35 (53) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 11 (12) | 3 (3)
Gastrointestinal - Other (Esophageal Obstruction) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (Hernia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Hemorrhage, CNS (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Upper GI NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 8 (10) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 7 (7) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 5 (5) | 0 (0) — (ANC <1.0 x 10e9/L)::Blood
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0 x 10e9/L)::Joint
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 5 (6) | 0 (0) — (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 2 (2) | 0 (0) — (ANC <1.0 x 10e9/L)::Skin (cellulitis)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 1 (1) — (ANC <1.0 x 10e9/L)::Small bowel NOS
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 2 (2) | 0 (0) — (ANC <1.0 x 10e9/L)::Upper airway NOS
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Rectum (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 5 (6) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Hip fracture) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 0 (0)
Neurology - Other (subdural hygroma) (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: cranial::CN VII Motor-face; Sensory-taste (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 (6) | 2 (2)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain - Other (Incision) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 4 (5)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain::Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 2 (2) | 0 (0)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Perforation, GI::Duodenum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perforation, GI::Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perforation, GI::Small bowel NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perforation, GI::Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Rash: dermatitis associated with radiation::Radiation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 0 (0)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | With EPOCH-R (Etoposide, Doxorubicin, Prednisone, Cyclophosphamide and Rituximab) (N=235) | EPOCH Alone (Etoposide, Doxorubicin, Prednisone, and Cyclophosphamide) (N=112)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 124 (210) | 19 (27)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 83 (121) | 12 (17)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 127 (231) | 15 (29)
Alkaline phosphatase (Metabolism and nutrition disorders) | 50 (72) | 14 (16)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 20 (24) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 62 (74) | 12 (14)
Amylase (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Anorexia (Gastrointestinal disorders) | 75 (122) | 18 (22)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Auditory/Ear - Other (decreased hearing) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 16 (34) | 2 (5)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 41 (62) | 7 (13)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 10 (17) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 60 (88) | 8 (8)
Cardiac General - Other (Fluid overload) (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Confusion (Nervous system disorders) | 6 (6) | 1 (2)
Constipation (Gastrointestinal disorders) | 146 (267) | 45 (65)
Constitutional Symptoms - Other (Intolerance to cold) (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 (81) | 10 (12)
Creatinine (Metabolism and nutrition disorders) | 26 (40) | 2 (2)
Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 24 (28) | 6 (6)
Dermatology/Skin - Other (Blisters-toes) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Cold sore) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 108 (184) | 43 (71)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 60 (84) | 12 (19)
Dry eye syndrome (Eye disorders) | 13 (13) | 5 (6)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 11 (12) | 4 (6)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 68 (94) | 16 (24)
Edema: limb (Blood and lymphatic system disorders) | 42 (52) | 11 (16)
Erectile dysfunction (Reproductive system and breast disorders) | 10 (17) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 11 (12) | 3 (5)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 2 (2) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 195 (417) | 78 (179)
Febrile neutropenia (Infections and infestations) | 41 (52) | 11 (11) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 77 (99) | 29 (45)
Fistula, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 12 (16) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 10 (11) | 2 (2)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal - Other (Bloating) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (Early satiety) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (Esophageal Stenosis) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal - Other (Hernia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 103 (194) | 19 (37)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 14 (17) | 4 (4)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 139 (154) | 80 (98)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 6 (7) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 55 (66) | 8 (9)
Hemoglobin (Blood and lymphatic system disorders) | 202 (580) | 36 (107)
Hemorrhage, GI::Anus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Hemorrhage, GI::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 14 (15) | 4 (4)
Hemorrhage, GI::Upper GI NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Varices (rectal) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage, GU::Urethra (Renal and urinary disorders) | 1 (3) | 0 (0)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 7 (7) | 2 (2)
Hemorrhage, GU::Vagina (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Hemorrhage, pulmonary/upper respiratory::Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 3 (3)
Hemorrhage, pulmonary/upper respiratory::Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (Ecchymosis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (Gluteal muscle;Compartment syndrome) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemorrhoids (Blood and lymphatic system disorders) | 7 (12) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 5 (5) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 (12) | 2 (2)
Hypertension (Cardiac disorders) | 5 (5) | 5 (5)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 32 (40) | 9 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 5 (5) | 9 (10)
Incontinence, urinary (Renal and urinary disorders) | 8 (8) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0 x 10e9/L)::Bladder (urinary)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 10 (10) | 4 (4) — (ANC <1.0 x 10e9/L)::Blood
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0 x 10e9/L)::External ear (otitis externa)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 5 (5) | 0 (0) — (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 12 (14) | 0 (0) — (ANC <1.0 x 10e9/L)::Mucosa
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 1 (1) — (ANC <1.0 x 10e9/L)::Pelvis NOS
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 3 (4) | 0 (0) — (ANC <1.0 x 10e9/L)::Rectum
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 3 (3) | 0 (0) — (ANC <1.0 x 10e9/L)::Skin (cellulites)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0 x 10e9/L)::Soft tissue NOS
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0 x 10e9/L)::Stomach
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0 x 10e9/L)::Upper airway NOS
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 4 (4) | 0 (0) — (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 2 (2) | 0 (0) — (ANC <1.0 x 10e9/L)::Vagina
Infection - Other (PAC; blood-yeast) (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (R axilla) (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (foot - tinea pedis) (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (fungal, tinea pedis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Abdomen NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 7 (7) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 1 (1) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Conjunctiva (Infections and infestations) | 2 (2) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::External ear (otitis externa) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lip/perioral (Infections and infestations) | 2 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Liver (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 7 (8) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Middle ear (otitis media) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Mucosa (Infections and infestations) | 13 (15) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nerve-peripheral (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nose (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Rectum (Infections and infestations) | 7 (7) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Salivary gland (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Scrotum (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 4 (4) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 3 (3) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Small bowel NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Ungual (nails) (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper aerodigestive NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 18 (19) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 8 (8) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vagina (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 2 (2) | 1 (1)
Infection with unknown ANC::Blood (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Conjunctiva (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC::Rectum (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Insomnia (Gastrointestinal disorders) | 53 (75) | 14 (17)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 7 (7) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 205 (1002) | 34 (142)
Lipase (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 185 (676) | 30 (100)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 54 (72) | 7 (12)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 57 (98) | 9 (16)
Memory impairment (Nervous system disorders) | 1 (1) | 3 (4)
Mood alteration::Agitation (Nervous system disorders) | 4 (4) | 3 (3)
Mood alteration::Anxiety (Nervous system disorders) | 20 (31) | 6 (9)
Mood alteration::Depression (Nervous system disorders) | 18 (32) | 5 (5)
Mucositis/stomatitis (clinical exam)::Large bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam)::Larynx (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 188 (520) | 88 (222)
Mucositis/stomatitis (clinical exam)::Stomach (Gastrointestinal disorders) | 3 (6) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 2 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 38 (45) | 10 (12)
Musculoskeletal/Soft Tissue - Other (Finger injury) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Hand cramps) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Hip fracture) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Spasms) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Sprain) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 24 (27) | 3 (3)
Nausea (Gastrointestinal disorders) | 155 (382) | 59 (123)
Neurology - Other (antonomic neuropathy) (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 29 (34) | 18 (23)
Neuropathy: sensory (Nervous system disorders) | 206 (301) | 88 (125)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 207 (917) | 39 (148)
Obstruction, GI::Small bowel NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ocular/Visual - Other (Red eye) (Eye disorders) | 1 (1) | 0 (0)
Ocular/Visual - Other (Uveitis) (Eye disorders) | 1 (1) | 0 (0)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 3 (3) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 43 (61) | 8 (9)
Pain - Other (Biopsy site) (General disorders) | 0 (0) | 1 (1)
Pain - Other (Epigastric) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pain - Other (Flank) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - Other (Groin) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain - Other (Lung) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain - Other (Ribs) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - Other (VAD site) (General disorders) | 1 (1) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 62 (79) | 22 (32)
Pain::Back (Musculoskeletal and connective tissue disorders) | 23 (34) | 8 (8)
Pain::Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 153 (373) | 24 (46)
Pain::Breast (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain::Buttock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 9 (11) | 2 (2)
Pain::Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 17 (19) | 2 (2)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pain::External ear (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 19 (21) | 7 (7)
Pain::Eye (Eye disorders) | 1 (1) | 1 (1)
Pain::Face (Skin and subcutaneous tissue disorders) | 10 (12) | 5 (6)
Pain::Head/headache (Nervous system disorders) | 99 (179) | 30 (45)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 54 (105) | 29 (41)
Pain::Larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain::Middle ear (Ear and labyrinth disorders) | 3 (4) | 0 (0)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 80 (125) | 29 (50)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 6 (6) | 0 (0)
Pain::Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain::Pain NOS (General disorders) | 2 (3) | 0 (0)
Pain::Pelvis (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Pain::Rectum (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (6)
Pain::Urethra (Renal and urinary disorders) | 8 (8) | 3 (3)
Pain::Vagina (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 17 (21) | 3 (4)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 9 (10) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 39 (64) | 5 (10)
Platelets (Blood and lymphatic system disorders) | 203 (841) | 36 (134)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 14 (19) | 7 (7)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 68 (130) | 9 (14)
Proctitis (Gastrointestinal disorders) | 6 (7) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 10 (14) | 1 (1)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 47 (56) | 17 (18)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7 (9) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal/Genitourinary - Other (Nocturia) (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal/Genitourinary - Other (dysuria) (Renal and urinary disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 22 (23) | 5 (10)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 19 (25) | 7 (12)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 87 (143) | 10 (13)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 3 (3) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 25 (32) | 4 (4)
Supraventricular and nodal arrhythmia::Supraventricular arrhythmia NOS (Cardiac disorders) | 2 (3) | 0 (0)
Sweating (diaphoresis) (General disorders) | 15 (17) | 5 (7)
Syncope (fainting) (Nervous system disorders) | 12 (12) | 0 (0)
Syndromes - Other (Akathisia) (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 76 (127) | 9 (12)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 24 (26) | 8 (9)
Tinnitus (Ear and labyrinth disorders) | 5 (6) | 1 (1)
Tumor lysis syndrome (General disorders) | 1 (1) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 12 (15) | 3 (4)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 3 (3) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vasovagal episode (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia::Ventricular arrhythmia NOS (Cardiac disorders) | 1 (1) | 0 (0)
Vision-blurred vision (Eye disorders) | 22 (28) | 5 (6)
Vision-flashing lights/floaters (Eye disorders) | 1 (1) | 0 (0)
Vision-photophobia (Eye disorders) | 4 (4) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 1 (1)
Vomiting (Gastrointestinal disorders) | 92 (147) | 31 (54)
Watery eye (epiphora, tearing) (Eye disorders) | 26 (27) | 3 (3)
Weight gain (General disorders) | 3 (3) | 0 (0)
Weight loss (General disorders) | 21 (22) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT00001337/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT00001337/ICF_001.pdf